CLINICAL TRIAL: NCT03459924
Title: Intraoperative Evaluation of Right Ventricular Function During Liver Transplantation: a Quantitative Analysis Using Transesophageal Echocardiography
Brief Title: Right Ventricular Function During Liver Transplantation as Assessed by Transesophageal Echocardiography.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, GLAUBER GOUVEA, Principal Investigator, Universidade Federal do Rio de Janeiro
Other Study IDs: 79763817.9.0000.5257
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Liver Transplant; Complications
Keywords: Right ventricular function; Liver transplantation; Transesophageal echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cirrhotic patients undergoing liver transplantation might develop acute transient right ventricular dysfunction, ranging from mild to severe form. More than two decades ago, a number of studies with pulmonary artery catheters looked at this particular issue with controversial results. However, the pulmonary artery catheter as a monitor for right ventricular function (RVF) has several limitations, while the echocardiogram is deemed to be more accurate in this regard. Therefore, we sought to evaluate the RVF with the transesophageal echocardiogram, and particularly whether the RVF significantly varies during this procedure.

DETAILED DESCRIPTION:
Evaluation of right ventricular function (RVF) during orthotopic liver transplantation (OLT) has been extensively reported with modified pulmonary artery catheters that measure the right ventricular ejection fraction. However, quantitative analysis of RVF using transesophageal echocardiography (TEE) are scarce in this setting.

Methods: Nineteen cirrhotic patients who underwent OLT from April-2012 to April-2013 will be studied. Analysis of echocardiogram-derived parameters routinely used to evaluate ventricular function will be done. In particular, the RVF was quantitatively assessed by two parameters derived from TEE: tricuspid annular plane systolic excursion (TAPSE) and right ventricular fractional area change (RVFAC). Exclusion criteria: pulmonary hypertension, fulminant hepatitis, age less than 18 or greater than 65 years old and cardiopulmonary diseases. All echocardiographic and hemodynamic data set have been collected at 5 stages during the procedure, according to Institutional Protocol: baseline, hepatectomy, anhepatic phase, post-reperfusion, and closure.

Statistical Analysis: One-way ANOVA for repeated measurements will be used if the data have normal distribution, otherwise Friedman test will be used. P<0.05 is to be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent orthotopic liver transplantation from april 2012 to april 2013.

Exclusion Criteria:

* Pulmonary hypertension (any type)
* Cardiopulmonary disease (eg: chronic obstructive pulmonary disease (COPD), valvular heart disease, ischemic heart disease)
* Fulminant hepatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cirrhotic patients who underwent a orthotopic liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Development of new right ventricular dysfunction during liver transplantation | Through study completion, after 1 year of data retrieval and analysis.
  Signs of right ventricular dysfunction as assessed by transesophageal echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Nubia V Figueiredo, MSc, PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis JE, Lichtor JL, Feinstein SB, Chung MR, Polk SL, Broelsch C, Emond J, Thistlethwaite JR, Roizen MF. Right heart dysfunction, pulmonary embolism, and paradoxical embolization during liver transplantation. A transesophageal two-dimensional echocardiographic study. Anesth Analg. 1989 Jun;68(6):777-82. PMID 2660629
- [Background] De Wolf AM, Begliomini B, Gasior TA, Kang Y, Pinsky MR. Right ventricular function during orthotopic liver transplantation. Anesth Analg. 1993 Mar;76(3):562-8. doi: 10.1213/00000539-199303000-00020. PMID 8452268
- [Background] Gouvea G, Diaz R, Auler L, Martinho JM. Evaluation of the right ventricular ejection fraction during orthotopic liver transplantation under propofol anaesthesia. Br J Anaesth. 2008 Aug;101(2):161-5. doi: 10.1093/bja/aen145. Epub 2008 Jun 4. PMID 18534974
- [Background] Gouvea G, Diaz R, Auler L, Toledo R, Martinho JM. Right ventricular ejection fraction during orthotopic liver transplantation: does anesthetic technique make a difference? J Crit Care. 2010 Dec;25(4):657.e1-6. doi: 10.1016/j.jcrc.2010.02.005. Epub 2010 Apr 8. PMID 20381292